CLINICAL TRIAL: NCT02689934
Title: Efficacy of Red Yeast Rice Based Nutraceutical (Monacolin K 10 mg/Dose) Plus Probiotic (Bifidobacterium Longum BB536 ®) in Patients With Moderate Hypercholesterolemia.
Brief Title: Efficacy of a Red Yeast Rice Based Nutraceutical Plus Probiotic in Patients With Moderate Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefarmaco OTC SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROBIOTICO - BB536
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; bifidobacterium longum BB536; red yeast rice; monacolin K; lactoflorene colesterolo
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind (subjects, investigators)

ARMS (2):
- Lactoflorene colesterolo (Experimental): Red Yeast Rice titrated in 10 mg monacolin K per daily dose plus Bifidobacterium longum 50 mg, powder form, 1 packet per day
  Interventions: Dietary Supplement: Lactoflorene colesterolo
- Placebo Lactoflorene colesterolo (Placebo Comparator): placebo, powder form, 1 packet per day
  Interventions: Dietary Supplement: Placebo lactoflorene colesterolo

INTERVENTIONS:
Dietary Supplement: Lactoflorene colesterolo — 1.8 g + 1.8 g once a day per os
  Arms: Lactoflorene colesterolo
Dietary Supplement: Placebo lactoflorene colesterolo — 1.8 g + 1.8 g once a day per os
  Arms: Placebo Lactoflorene colesterolo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel study to evaluate the efficacy of a red yeast rice based nutraceutical (monacolin K 10 mg/dose) plus probiotic (Bifidobacterium longum BB536 ®), versus placebo, in patients with moderate hypercholesterolemia, in terms of improvement of the lipid profile and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ men or women ≤ 70
* men or female. Female must be postmenopausal or surgically sterile
* 130 mg/dl ≤ LDL-C ≤ 200 mg/dl
* patients in primary cardiovascular prevention

Exclusion Criteria:

* pregnancy and lactating
* patients with chronic diseases
* patients with serious hepatic diseases
* patients with serious renal diseases
* patients with thyroid diseases
* diabetes mellitus or glycemia >126 mg/dl
* uncontrolled or severe hypertension
* obesity(BMI>30)
* smoking status
* drug or nutraceutical that can interfere with the experimental treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02-21 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Percent Change in LDL-C From Baseline | 12 weeks
  Percent change from baseline in LDL-C after 12 weeks of treatment in patients with moderate hypercholesterolemia

SECONDARY OUTCOMES:
Safety and tolerability of Lactoflorene colesterolo (Incidence of treatment-related adverse events) | 12 weeks
  Incidence of treatment-related adverse events
Changes in Other Lipids (non HDL-C, TG, HDL-C) and Apolipoproteins | 12 weeks
Changes in Vital Signs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana G Mombelli, MD, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda Cà Granda
Locations (1):
- Centro Dislipidemie Dip. Cardiotoracovasc ASST Grande Ospedale Metropolitano Niguarda Cà Granda, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruscica M, Pavanello C, Gandini S, Macchi C, Botta M, Dall'Orto D, Del Puppo M, Bertolotti M, Bosisio R, Mombelli G, Sirtori CR, Calabresi L, Magni P. Nutraceutical approach for the management of cardiovascular risk - a combination containing the probiotic Bifidobacterium longum BB536 and red yeast rice extract: results from a randomized, double-blind, placebo-controlled study. Nutr J. 2019 Feb 22;18(1):13. doi: 10.1186/s12937-019-0438-2. PMID 30795775
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/30795775